CLINICAL TRIAL: NCT00183807
Title: A Phase II Study of Irinotecan (Camptosar), Cisplatin and Celebrex in Patients With Metastatic or Unresectable Esophageal Cancer
Brief Title: A Study of Irinotecan, Cisplatin and Celebrex in Patients With Metastatic or Unresectable Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3E-02-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Irinotecan; Cisplatin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan, cisplatin, celecoxib

SUMMARY:
This study is for patients with cancer of the esophagus. This study uses the drugs irinotecan, cisplatin and celecoxib. Irinotecan (also known as CPT-11) was recently approved by the U.S. Food and Drug Administration (FDA) for use in colon cancer, but has not been approved by the FDA for use in the treatment of cancers of the esophagus. Cisplatin is a drug that is commonly used to treat patients with cancer of the esophagus. We are combining these two chemotherapy drugs with a drug called Celebrex. Celebrex (also called Celecoxib) is an oral medication that is approved by the FDA for pain in the treatment of arthritis. There is some information to suggest that this drug may have anti-cancer activity. In prior studies combining irinotecan and cisplatin, tumors of the esophagus have been shown to shrink. We are adding Celebrex to these drugs to see if it makes the drugs work better to shrink cancer or cause fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented unresectable or metastatic esophageal cancer and histologic confirmation of the diagnosis with tumor. To be unresectable a patient must have been examined by a surgeon and declared unresectable.
* Tissue from tumor must be available. This may be paraffin embedded tissue from previous biopsy/resection or if it is not available, a repeat biopsy must be performed.
* Patients must agree to have a sample 20 cc drawn in addition to routine labs with each cycle of chemotherapy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan. If prior radiation therapy was administered, measurable disease must be outside the radiation field.
* Patients may have received prior adjuvant chemotherapy; this must have been completed at least 6 months prior to the initiation of therapy for metastatic disease.
* Patients must have a Zubrod performance status of 0-2.
* Patients must have a predicted life expectancy of at least 12 weeks.
* Patients must have a pre-treatment granulocyte count (i.e., segmented neutrophils + bands) of >1,500/mm3, a hemoglobin level of greater than or equal to9.0 gm/dl, and a platelet count of >100,000/mm3.
* Patients must have adequate renal function as documented by

  1) creatinine less than or equal to 1.5 X institutional upper limit of normal OR 2) creatinine clearance > 60 mL/min as calculated with
* Patients must have adequate hepatic function as documented by a serum bilirubin less than or equal to 2x the institutional upper limit of normal, regardless of whether patients have liver involvement secondary to tumor. Aspartate transaminase (SGOT) must be less than or equal to 3x institutional upper limit of normal, unless the liver is involved with tumor, in which case the aspartate transaminase must be less than or equal to 5x institutional upper limit of normal.
* No major surgery within 1 month of starting study drug.

Exclusion Criteria:

* Patients who have received prior therapy with CPT-11 or cisplatin as adjuvant therapy less than 12 months prior to initiation of therapy for metastatic disease. All other adjuvant chemotherapy must have been completed at least 6 months prior to entry onto trial.
* Prior treatment with celebrex, that is if patients are currently using celebrex on a regular basis for the treatment of other disorders, i.e arthritis, etc.
* Patients who have received prior treatment for metastatic or unresectable disease
* Patients taking full-dose NSAIDs, including aspirin, regularly for any reason (e.g., arthritis, history of TIA or myocardial infarction). Patients taking cardiac preventive dose ASA (<81mg daily) are eligible. Patients should stop taking any other NSAIDs 14 days prior to receiving first dose of Celecoxib.
* Patients may not have a history of an allergy to sulfonamide drugs.
* Patients may not have active peptic ulcer disease or other contraindications to chronic NSAID use or aspirin use.
* Patients may not have known lactose intolerance.
* Patients with any active or uncontrolled infection, including known HIV infection
* Patients with psychiatric disorders that would interfere with consent or follow-up
* Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis
* Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other anti-epileptic prophylaxis are ineligible.
* Patients with uncontrolled diabetes mellitus, defined as random blood sugar greater than or equal to 200 mg/dl.
* Patients with any other severe concurrent disease, which in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-10; Primary Completion 2006-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To assess the time to progression of CPT-11 and cisplatin in combination with celebrex in patients with metastatic or unresectable carcinoma of the esophagus

SECONDARY OUTCOMES:
To assess response rate and overall survival in these patients.
To assess the toxicity of this regimen.
To identify molecular correlates of response and survival (gene expression and genomic polymorphism of enzymes involved in drug metabolism, DNA repair, apoptosis)
To evaluate the effects of celebrex on a variety of histological and molecular biomarkers of angiogenesis, including in vitro activity assays on endothelial cell proliferation, migration and invasion.

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C./ Norris Comprehensive Cancer Center
Locations (1):
- U.S.C. / Norris Comprehensive Cancer Center, Los Angeles, California, United States